CLINICAL TRIAL: NCT03697200
Title: Auricular Point Acupressure to Self-Manage Chronic Pain or Aromatase Inhibitor Musculoskeletal Symptoms in Breast Cancer Survivors: Effectiveness and Scientific Underpinnings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00158622
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Aromatase Inhibitor; Musculoskeletal Symptoms; Postmenopausal Breast Cancer Survivors
Keywords: Breast Cancer Survivors; Aromatase Inhibitor; Ecological Momentary Assessment; Musculoskeletal Symptoms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auricular Point Acupressure (APA) (Active Comparator): Patients with active points related to Aromatase Inhibitor Musculoskeletal Symptoms (AIMSS). The points for AIMSS include (1) points corresponding to body pain location and (2) three points known for alleviating stress and pain (i.e., shenmen, sympathetic, and nervous subcortex)
  Interventions: Other: APA
- Sham APA control (Sham Comparator): The same procedure of APA will be applied but the tapes/seeds will be placed on different points (points not related to AIMSS). Participants in the Sham APA Control will receive APA on the five ear points comprising mouth, stomach, duodenum, internal ear, and tonsils. These points are chosen for the Sham APA Control for two reasons: First, they are distinct from the zones of the ear (and the points therein) associated with AIMSS and correspond to body regions in which BCS (Breast Cancer Survivors) are usually pain-free; second, they are equivalent in number to those points used in the APA treatment group and no negative impacts have been observed among these points in our pilot study.
  Interventions: Other: Sham APA control
- Education Control (Other): Participants in the Education Control will receive four, 15-minute weekly individual sessions in which the scheduling and duration of interaction with the study staff are identical to the APA and Sham interventions. Educational sessions are intended to reflect usual standard medical care per guidelines from the American Society of Clinical Oncology (ASCO), while also meeting the needs of trial participation, including (1) the knowledge of hormonal therapy and side effects; (2) assessment and management of physical long-term and late effects; (3) assessment and management of psychological long-term and late effects; and (4) dietary (developed by Co-I, van Londen) and physical activity in Breast Cancer Survivors (BCS) (developed by Co-I, Stearns). These materials have been used by the research team, and clinical practice. Materials will be tailored so that they can be delivered within 15 minutes for each session.
  Interventions: Other: Education control

INTERVENTIONS:
Other: APA — Light touch using vaccaria seeds on specific points of the ear
  Arms: Auricular Point Acupressure (APA)
Other: Sham APA control — Light touch using vaccaria seeds on different points of the ear (compared to the APA group).
  Arms: Sham APA control
Other: Education control — Participants in the Education Control will receive four, 15-minute weekly individual sessions in which the scheduling and duration of interaction with the study staff are identical to the APA and Sham interventions. Materials will be tailored so that they can be delivered within 15 minutes for each session
  Arms: Education Control

SUMMARY:
Aromatase inhibitor therapy has become a standard adjuvant endocrine therapy for postmenopausal women with hormone receptor-positive breast cancer. Up to 50% of postmenopausal breast cancer survivors exhibit significant aromatase inhibitor musculoskeletal symptoms, defined as severe joint pain and stiffness. Aromatase inhibitor musculoskeletal symptoms in turn has a negative effect on the women's physical function and quality of life, leading to discontinued aromatase inhibitor therapy and causing significant social and economic burden. Given aromatase inhibitor musculoskeletal symptoms' profound effects, the management of aromatase inhibitor musculoskeletal symptoms is an essential component in cancer care.

The investigators propose to test auricular point acupressure- -an innovative, non-invasive, nonpharmacologic, and low-cost intervention- -to manage aromatase inhibitor musculoskeletal symptoms in breast cancer survivors. Auricular point acupressure applies an acupuncture-like stimulation to ear acupoints without using a needle (i.e., seeds are taped to the acupoints) to treat illness/symptoms. Auricular point acupressure is particularly well suited for current challenges of unmet aromatase inhibitor musculoskeletal symptoms management. The investigators propose a randomized controlled trial to (1) determine the efficacy of auricular point acupressure in relieving aromatase inhibitor musculoskeletal symptoms, and (2) examine the inflammatory signaling of auricular point acupressure effects in breast cancer survivors treated with aromatase inhibitor. The investigators will also measure psychological, behavioral, personal, and social factors that may moderate or mediate the effects of auricular point acupressure. The investigators also believe inflammatory cytokines may partially explain the mechanism of action of auricular point acupressure for improved aromatase inhibitor musculoskeletal symptoms and physical function, and plan to measure these.

This study will identify a novel approach to manage aromatase inhibitor musculoskeletal symptoms in postmenopausal breast cancer survivors, with minimal side effects. If successful, the paradigm of pain management will shift from a traditional medical model to a larger integrative medicine and patient-management paradigm to avoid unnecessary evolution towards prolonged disability.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of Breast Cancer (non-metastatic) before entering into postmenopausal age
* Currently receiving AIs (anastrazole, letrozole, exemestane) per chart documentation for at least 2 months (the peak onset of AIMSS is 1.6 months).
* Able to read and write English
* Have joint pain attributable to AI-or had pre-existing joint pain that worsened after the initiation of AIs-and had worst joint pain rated as 4 or more on a 0-10 numeric rating scale in the previous week
* Are willing to commit to weekly study visits for 4 weeks during the intervention and monthly follow-up visits for 3 months (up to 4 months)
* Able to apply pressure to the seeds taped to the ears

Exclusion Criteria:

* Metastatic breast cancer
* Completed cytotoxic chemotherapy or radiation therapy less than 4 weeks prior to enrollment (because chemotherapy and radiation therapy can cause temporary exacerbation of joint symptoms that typically resolve spontaneously)
* Bone fracture/surgery of an affiliated extremity during the preceding 6 months
* Current use of corticosteroids or narcotics
* Ear skin disease
* Allergy to the tape used for this study
* Having had previous auricular therapy (because they would be unable to be blinded for the study)
* Having been hospitalized for mental health reasons within the last 3 months
* Piercings on the ear points for treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with a history of Breast Cancer (non-metastatic) before entering into postmenopausal age
Enrollment: 102 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity as assessed by the Brief Pain Inventory-short form | Baseline, pre- Intervention (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), and 3-month (20 weeks)
  The Brief Pain Inventory-short form (BPI-sf) questionnaire includes assessment of pain location and multiple aspects of severity of pain, numbness, tingling, and stiffness, including worst, least, average pain, and present, as well as the interference with daily activities. The Brief Pain Inventory-short form (BPI-sf) has a total score ranging from 0 to 10 with higher scores indicating more pain.
Change in Physical Function as assessed by the Western Ontario and McMaster Osteoarthritis Index | Baseline, pre- Intervention (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), and 3-month (20 weeks)
  The Western Ontario and McMaster Osteoarthritis Index (WOMAC) consists of 24 items divided into 3 subscales:
  * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing
  * Stiffness (2 items): after first waking and later in the day
  * Physical Function (17 items): stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties.
  The WOMAC score range from 0 to 96. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change in Physical disability as assessed by the QuickDASH | Baseline, pre- Intervention (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), and 3-month (20 weeks)
  QuickDASH outcome measure is used. At least 10 of the 11 items must be completed for a score to be calculated. The assigned values for all completed responses are simply summed and averaged, producing a score out of five. The value is then transformed to score out of 100. The score range will be 0 to 100. Higher score indicating greater disability.
Change in Physical Strength as assessed by Handgrip | Baseline, pre- Intervention (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), and 3-month (20 weeks)
  Handgrip strength is a simple and commonly used test of a person's general strength level. There is a simple norm table which is categorized with age is used to measure the strength.

SECONDARY OUTCOMES:
Change in medication use adherence as assessed by the Ecological Momentary Assessment | Baseline, pre- Intervention (4 weeks), post-intervention (8 weeks), one-month (12 weeks), 2-month (16 weeks), and 3-month (20 weeks)
  Analgesic use and Aromatase Inhibitor (AI) adherence will be included in the Ecological Momentary Assessment (EMA) diary during intervention and medications will be checked at study visits at follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Chao H Yeh, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No